CLINICAL TRIAL: NCT07138599
Title: Training Healthcare Professionals in an Artificial Intelligence Based Virtual Reality Extracorporeal Membrane Oxygenation Simulator Versus Conventional Video Training; a Multicentre Feasibility Study and Randomised Controlled Trial
Brief Title: Virtual Reality Training for ECMO Circuit Checks
Acronym: HEALTH-ECMO-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Edris Mahtab, MD PhD, Cardiothoracic Surgeon & PI, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MEC-2023-0666; LUMC Fellowship Grant 2023 (Other Grant/Funding Number: Leiden University Medical Center)
Record Dates: First submitted 2025-07-30; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: ECMO; Training Effectiveness; Education Nursing; Educational Intervention; Virtual Reality; Simulation Based Medical Education; Simulation Training
Keywords: ECMO; Virtual Reality; Simulation; Medical Education; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional EMCO Circuit Check Training (Active Comparator): Participants allocated to the conventional video training arm will view a narrated video recording in which two certified perfusionists give a standard educational talk and demonstration that they provide when educating new intensive care unit staff and perfusionists-in-training. The identical eleven step circuit check on a primed wet circuit matches the equipment used for outcome assessment. The video will be presented on a laptop with headphones in a quiet room with minimal distractors, after which learners may asks questions or clarification from the study coordinator prior to the beginning of the assessment.
  Interventions: Other: Instructional Video of Certified Perfusionists on Performing a Circuit Check
- Virtual Reality ECMO Circuit Check Simulation Training Novice Group (Experimental): Novice participants assigned to the Virtual Reality Simulation arm will undergo a fifteen minute individual session delivered on a Meta Quest 3 headset that simulates a fully interactive extracorporeal membrane oxygenation circuit. The scenario will guide each learner through the eleven prescribed safety checks while allowing manipulation of circuit components and providing immediate audio visual feedback. No further instruction will precede the subsequent live assessment. This arm then undergoes the physical assessment on a physical ECMO practice circuit.
  Interventions: Device: Virtual Reality ECMO Simulation Training
- Experimental: Virtual Reality ECMO Circuit Check Simulation Training Expert Group (Other): Expert participants assigned to the Virtual Reality Simulation arm will undergo a fifteen minute individual session delivered on a Meta Quest 3 headset that simulates a fully interactive extracorporeal membrane oxygenation circuit. The scenario will guide each learner through the eleven prescribed safety checks while allowing manipulation of circuit components and providing immediate audio visual feedback. This arm is then asked to complete a questionnaire regarding the relevance of each of the steps in the circuit check to investigate the content validity. Participants then fill out a USE questionnaire with the purpose of demonstrating face validity.
  Interventions: Device: Virtual Reality ECMO Simulation Training

INTERVENTIONS:
Device: Virtual Reality ECMO Simulation Training — The intervention is a virtual reality simulation of an ECMO system, whereby the user is guided through the steps of how to perform an 11 step ECMO circuit check, and specific indicators of abnormal functioning are highlighted. The simulation is produced in Unreal Engine 4.23, and it simulates a virtual ICU and a virtual patient.
  Other Names: VR ECMO-sim; Virtual Reality Extracorporeal Membrane Oxygenator
  Arms: Experimental: Virtual Reality ECMO Circuit Check Simulation Training Expert Group; Virtual Reality ECMO Circuit Check Simulation Training Novice Group
Other: Instructional Video of Certified Perfusionists on Performing a Circuit Check — This intervention is a seven minute narrated high definition video in which a two certified perfusionist describe how to perform the identical eleven step circuit check on a primed Cardiohelp circuit, what to look for in terms of pathology or abnormal function, and . Participants will view the clip once on a laptop with headphones in a quiet room and may ask questions or receive clarification from the study coordinator, and this will be demonstrated on the physical ECMO machine and/or circuit present. The video conveys the checklist at reduced speed and explaining the purpose of each step and has been reviewed by the expert panel for accuracy and completeness.
  Other Names: Conventional Training
  Arms: Conventional EMCO Circuit Check Training

SUMMARY:
Purpose of the Study:

This investigation will examine whether a brief session with an immersive virtual-reality headset can prepare critical-care nurses to carry out an eleven-step extracorporeal membrane oxygenation circuit check as accurately and as quickly as the standard narrated training video that clinicians normally watch at the bedside.

Who Will Take Part:

Two groups of volunteers will be enrolled. Eight senior clinicians who already have at least five years of extracorporeal membrane oxygenator experience will test the simulator so that investigators can confirm its realism and educational relevance. In a separate arm, forty-four intensive-care or cardiothoracic nurses with no prior ECMO training or ECMO patient care experience.

How Participants Will Be Assigned:

Nurses will be allocated by computer in a one-to-one ratio either to the virtual-reality session or to the video. Because the assignment sequence will be generated in advance and concealed inside a secure web form, neither facilitators nor learners will be able to predict the next allocation. The two examiners who will judge each live circuit check will not be told which training each nurse received.

What Will Happen During the Study:

Experts will first complete a single virtual-reality scenario that guides them through the eleven checks on a simulated circuit. Immediately afterward they will rate the experience with the standard Usefulness Satisfaction and Ease-of-Use questionnaire.

Nurses will then receive their assigned training. The virtual-reality group will spend fifteen minutes practising the checklist inside a standalone headset, while the video group will watch a seven-minute narrated recording that mirrors the usual bedside demonstration.

After training every nurse will complete a real circuit check on a primed wet circuit. A blinded examiner will watch the procedure, score each of the eleven checklist items, and time the task from start to finish.

Measurements the Researchers Will Use:

For nurses the primary measurements will be the number of checklist items missed and the total time needed to finish the procedure. For experts the main measurements will be their ratings of realism, usefulness, and ease of use. Investigators will also explore the link between the kind of training received and performance during the wet-lab task to confirm whether the simulator provides valid learning.

Where and For How Long the Study Will Run The investigation will take place at two university medical centres in the Netherlands. Each participant's involvement will last no longer than one day, and the entire study is expected to be completed within twelve months of first enrolment.

How Many People Will Take Part and Why:

Statistical calculations show that twenty-two nurses in each arm will give more than eighty-five per cent power to detect one missed checklist item between groups when the type-one error rate is five per cent. Allowing for potential withdrawals, forty-four novices and eight experts will be recruited.

Why the Study Design Matters:

By combining an expert validation phase with a randomised, assessor-blinded trial in novices, the study will determine both the realism of the virtual-reality simulator and its ability to improve real-world performance.

DETAILED DESCRIPTION:
This investigation will be a prospective multicentre study that integrates a preparatory validation phase with a concealed-allocation randomised controlled trial. Its central purpose will be to determine whether an immersive virtual reality module can reproduce the realism of a wet laboratory and transfer measurable skill to novices who must perform an eleven-step extracorporeal membrane oxygenation circuit check. The clinical need for scalable, high-fidelity training, together with encouraging early feasibility work in related simulators, provides the scientific rationale for this protocol .

Two Dutch university hospitals will serve as recruiting sites. In phase one eight consultant intensivists or senior perfusionists with at least five years of extracorporeal experience will complete a single scenario inside the Virtual-Reality Extracorporeal Membrane Oxygenation Simulator and will then answer the nineteen-item Usefulness Satisfaction and Ease-of-Use questionnaire. Their judgments will supply evidence for face and content validity according to the Messick framework.

Phase two will enrol forty-four intensive-care or cardiothoracic nurses who have never operated the Cardiohelp platform. A computer-generated list prepared with Research Randomizer will assign them in a one-to-one ratio either to a VR training session, or to a seven minute narrated training video that mirrors conventional bedside teaching. Allocation will be concealed by an automated Microsoft Forms workflow so that trainers cannot foresee the next assignment; video assessors who will later rate performance will remain masked to group allocation.

The virtual reality module will be delivered on stand-alone Meta Quest headsets, with a simulation produced with Unreal Engine. The control video will be shown on a laptop with headphones and will depict licensed perfusionists demonstrating the identical checklist in real time, after which learners may ask questions from the coordinator, who will answer them using the physical ECMO circuit that is present.

Immediately after their assigned training every novice will complete an physical circuit check on a primed wet circuit with a Cardiohelp console. This assessment is filmed and later assessed by an examiner, blinded to allocation, who will score the procedure from video using an eleven-item checklist validated by the expert panel and will record total completion time. The assessment encounter itself will constitute an external criterion that will permit concurrent validity testing .

All questionnaire data will be captured through encrypted Microsoft Forms and stored in SharePoint, where automatic linkage to study identifiers will occur. Raw video files will be retained on a secure institutional drive with mirrored backup in SharePoint. After database lock, a de-identified archive will be created and preserved for ten years under Erasmus MC and Leiden UMC governance .

Power analysis based on a projected mean difference of 1 checklist error and a standard deviation of 1.1 showed that 16 novices per arm will provide at least eighty percent power at the 5% significance level; the same computation justified recruiting eight experts for the validation phase .

Primary analyses will follow an intention-to-treat principle. Continuous variables will first undergo Shapiro-Wilk testing; normally distributed outcomes will be compared with independent samples t tests, whereas non-normal data will use the Mann-Whitney U statistic. Categorical data will be analysed with Chi squared or Fisher exact tests as appropriate. Confounding will be explored with analysis of covariance when indicated, and significance will be declared at p<0.05.

Quality assurance will rest on several safeguards. Assessors will complete calibration sessions before scoring begins, database logic checks in Microsoft Forms will limit data entry errors, and the coordinating centres will perform audits of consent forms, randomisation logs and source videos against electronic records.

Risks are considered minimal. A small proportion of participants may experience transient nausea while wearing the headset, but symptoms usually resolve promptly once the display is removed; no other adverse effects are foreseen .

The study will adhere to the Declaration of Helsinki and GDPR legislation. Written informed consent will be obtained from every participant, and ethical approval has already been granted by the boards of both participating centres. Upon completion, the anonymised dataset and accompanying data dictionary will be deposited in Zenodo, enabling independent verification and secondary analyses

By pairing validity evidence with an assessor-blinded randomised comparison, this protocol will clarify whether an inexpensive head-mounted display can deliver training that is realistic, comprehensive and transferable to the bedside, setting a template for future immersive-simulation research in extracorporeal membrane oxygenator support.

ELIGIBILITY:
Expert Cohort

Inclusion Criteria:

I. Licensed consultant intensivist or certified clinical perfusionist with ≥ 5 years ECMO experience II. Currently employed at one of the participating centres III. Provides written informed consent

Exclusion Criteria:

I. History of severe motion-sickness, vertigo, seizure disorder, or uncorrected visual/vestibular impairment that precludes safe VR use

Novice Cohort

Inclusion Criteria:

I. Registered ICU or cardiothoracic-surgery nurse with no experience with the Cardiohelp ECMO system II. Age ≥ 18 years III. Able to understand written and spoken Dutch IV. Provides written informed consent

Exclusion Criteria:

I. Any formal Cardiohelp ECMO course, wet-lab, or VR ECMO session completed before enrolment II. As per experts: severe motion-sickness, seizure disorder, uncorrected visual/vestibular impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Missed Items During the ECMO Circuit Check | Assessment performed immediately after the conclusion of the VR or conventional training.
  For every participant, the eleven mandatory steps will be scored as correct or incorrect by an independent assessors who are masked to training allocation and who review the video recording of the live assessment. The total count of items marked incorrect will be recorded for each participant. The mean number of missed items in each study arm will be used as the analytic metric. Lower counts indicate better performance.
Time Needed to Complete the Eleven Step ECMO Circuit Check | Assessment performed immediately after the conclusion of the VR or conventional training.
  For every participant, the interval in seconds from first contact with the circuit to verbal declaration of completion will be measured and verified against the video timestamp by the independent assessors who are masked to training allocation. The mean completion time in seconds will be compared between study arms. Shorter times indicate better performance.

SECONDARY OUTCOMES:
Proportion of Participants Requiring Assistance During the Circuit Check | Assessment performed immediately after the conclusion of the VR or conventional training.
  During the live assessment each assessor will note whether the participant requests or receives any external help. The proportion of participants who require assistance will be calculated for each study arm.
VR Simulator Face Validity Score (USE Questionnaire Total) | Questionnaire filled in immediately after the completion of the VR simulation.
  Immediately after completing the virtual reality scenario each expert will complete the nineteen item Usefulness Satisfaction and Ease of Use Questionnaire. Item scores range from one to five and are summed to give a total from nineteen to ninety five, with higher totals indicating greater perceived realism, usefulness and ease of use. The mean total score across experts will constitute the outcome metric.
Simulator Content Validity Index | Questionnaire filled in by expert cohort immediately after the completion of the VR simulation.
  Experts will rate the relevance of each checklist element on a four point ordinal scale. The scale content validity index will be calculated as the proportion of items that receive a relevance rating of three or four. Values above 0.80 are interpreted as good content coverage.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus MC University Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on Zenodo for reuse.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be hosted for a minimum of 20 years through the Zenodo platform.
Access Criteria: A DOI link will be made available in the publication to the data, and requests to access the data can be made through the Zenodo platform.

REFERENCES:
- [Background] Mahtab EAF, Max SA, Braun J, Regeer MV, Kaufman B, Dunning J, Bibleraaj B, Andreas M, Rodriguez Lecoq R, Klinceva M, Rosalia R, Lorusso R, Bruining N, Egorova AD. Developing a Systematic Approach for the Implementation of Medical Extended Reality Learning Modules in Cardiothoracic Health Care: Recommendations From an International Expert Group. JACC Adv. 2025 Feb 26;4(3):101633. doi: 10.1016/j.jacadv.2025.101633. Online ahead of print. PMID 40147055
- [Background] Sadeghi AH, Peek JJ, Max SA, Smit LL, Martina BG, Rosalia RA, Bakhuis W, Bogers AJ, Mahtab EA. Virtual Reality Simulation Training for Cardiopulmonary Resuscitation After Cardiac Surgery: Face and Content Validity Study. JMIR Serious Games. 2022 Mar 2;10(1):e30456. doi: 10.2196/30456. PMID 35234652
- [Background] Peek JJ, Max SA, Bakhuis W, Huig IC, Rosalia RA, Sadeghi AH, Mahtab EAF. Virtual Reality Simulator versus Conventional Advanced Life Support Training for Cardiopulmonary Resuscitation Post-Cardiac Surgery: A Randomized Controlled Trial. J Cardiovasc Dev Dis. 2023 Feb 4;10(2):67. doi: 10.3390/jcdd10020067. PMID 36826563
- [Background] Babar ZUD, Max SA, Martina BG, Rosalia RA, Peek JJ, van Dijk A, Sadeghi AH, Mahtab EAF. Virtual reality simulation as a training tool for perfusionists in extracorporeal circulation: Establishing face and content validity. JTCVS Tech. 2023 Jun 20;21:135-148. doi: 10.1016/j.xjtc.2023.06.004. eCollection 2023 Oct. PMID 37854847

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT07138599/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Document for Novices (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT07138599/ICF_001.pdf
  • Informed Consent Form: Informed Consent Document for Experts (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT07138599/ICF_002.pdf